CLINICAL TRIAL: NCT05421533
Title: A Global Prospective observationAl Study of Real-worlD managemEnt of patieNts With atrIal fibrillAtion at High Risk of Stroke (GARDENIA)
Brief Title: Study in Atrial Fibrillation (AF) Patients at High Risk of Stroke
Acronym: GARDENIA
Status: Terminated | Type: Observational
Why Stopped: Concentration of resources on Phase 3 studies
Sponsor: Anthos Therapeutics, Inc. (Industry)
Collaborators: CYTE Global (Network)
Responsible Party: Sponsor
Other Study IDs: ANT-401
Record Dates: First submitted 2022-06-06; First posted 2022-06-16 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation
Keywords: Observational Study; Real-World Evidence; Atrial Fibrillation; Stroke; Bleeding; Systemic Thromboembolic Event
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The GARDENIA registry will collect real-world clinical data on the anticoagulant strategies in patients with AF at elevated risk of stroke but also elevated risk of bleeding.

DETAILED DESCRIPTION:
The GARDENIA registry will collect real-world clinical data on the utilization of oral anticoagulants in patients with atrial fibrillation (AF) at elevated risk of stroke. Patients with AF who meet 1 or more of the following criteria will be recruited: advanced age, renal dysfunction, the need for concomitant antiplatelet use, or otherwise judged to be at a higher risk of bleeding. Patients with these criteria are frequently not treated with currently approved oral anticoagulants or they are 'undertreated' based on the use of non-recommended doses of anticoagulants. These patients will be described with regards to baseline demographics and characteristics with particular attention focused on physician and patient factors that may play a role in the under use of guideline-recommended anticoagulation therapy for stroke prevention in patients with AF. Patients in the registry will also be followed to determine the rates of discontinuation/switching of their anticoagulation therapy, incidence of major adverse cardiovascular events and clinically relevant outcome events related to the selection of their anticoagulation therapy. The collected real-world data will be used to inform future studies of patients with AF at elevated risk of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient, or legally authorized representative, must be obtained before any assessment is performed
* Patients with diagnosed AF or atrial flutter(documented on an electrocardiogram or monitor recording)
* CHA2DS2-VASc score ≥2 excluding female as a factor
* Judged by the investigator to be at increased risk of bleeding because of at least 1 of the following:

  * Age ≥70on the day of informed consent
  * Reduced renal function (creatinine clearance <30mL/min by Cockcroft-Gault)
  * Chronic use of NSAIDs or antiplatelet agents
  * Any other condition associated with increased risk such as a prior history of major or clinically relevant nonmajor bleeding, increased fall risk, or frailty
* Patients who are not treated with oral anticoagulants (only applies to the initial feasibility cohort)

Exclusion Criteria:

* Mechanical heart valve or valve disease that is expected to require valve replacement intervention (surgical or invasive) during the course of the registry study
* AF due to a reversible cause (eg, cardiac surgery, pulmonary embolism, untreated hyperthyroidism, ethanol use)
* Clinical unstable or active endocarditis or endovascular infection
* Patients with a medical condition other than AF for which chronic use of an oral anticoagulant is indicated
* History of left atrial appendage closure or removal
* Life expectancy <1 year at the time of enrollment as assessed by the investigator
* Any medical or psychiatric condition which in the judgment of the Investigator may preclude patients from complying with study requirements for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AF at elevated risk of stroke with advanced age, renal dysfunction, the need for concomitant antiplatelet use, or otherwise judged to be at increased risk of bleeding. Initial feasibility cohort will recruit approximately 1500 patients with AF who are not currently treated with oral anticoagulants at baseline before opening the study to patients with AF regardless of antithrombotic strategy.
Sampling Method: Non-Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Distribution of characteristics of patients with AF, including reasons anticoagulation is not used | 24 Months
  Information collected from physicians will provide the clinical reasons for treatment or nontreatment with OACs as assessed by the treating physicians
Bleeding | 24 Months
  Number of all bleeding events in patients with AF who are treated with guideline recommended doses of oral anticoagulants for stroke prevention versus those who are not
Stroke and systemic embolic events | 24 Months
  Number of stroke and systemic embolic events in patients with AF who are treated with guideline recommended doses of oral anticoagulants for stroke prevention versus those who are not

CONTACTS AND LOCATIONS:
Locations (94):
- United States (9):
  - Anthos Investigate Site, Fullerton, California
  - Anthos Investigate Site, Boca Raton, Florida
  - Anthos Investigative Site, Homestead, Florida
  - Anthos Investigate Site, Atlanta, Georgia
  - Anthos Investigate Site, Marietta, Georgia
  - Anthos Investigative Site, Lanham, Maryland
  - Anthos Investigate Site, Detroit, Michigan
  - Anthos Investigate Site, Cary, North Carolina
  - Anthos Investigate Site, Tomball, Texas
- Argentina (17):
  - Anthos Investigate Site, Caba, Buenos Aires
  - Anthos Investigate Site, Coronel Suárez, Buenos Aires
  - Anthos Investigate Site, La Plata, Buenos Aires
  - Anthos Investigate Site, Quilmes, Buenos Aires
  - Anthos Investigate Site, Ramos Mejía, Buenos Aires
  - Anthos Investigate Site, San Nicolás de los Arroyos, Buenos Aires
  - Anthos Investigate Site, Buenos Aires, Buenos Aires F.D.
  - Anthos Investigate Site, Córdoba, Córdoba Province
  - Anthos Investigate Site, Esperanza, Santa Fe Province
  - Anthos Investigate Site, Granadero Baigorria, Santa Fe Province
  - Anthos Investigate Site, Rosario, Santa Fe Province
  - Anthos Investigate Site, San Miguel de Tucumán, Tucumán Province
  - Anthos Investigate Site, Corrientes
  - Anthos Investigate Site, Córdoba
  - Anthos Investigate Site, Salta
  - Anthos Investigate Site, San Luis
  - Anthos Investigate Site, Santa Fe
- Brazil (9):
  - Anthos Investigate Site, Colatina, Espírito Santo
  - Anthos Investigate Site, Campo Grande, Mato Grosso do Sul
  - Anthos Investigate Site, Belo Horizonte, Minas Gerais
  - Anthos Investigate Site, Campina Grande do Sul, Paraná
  - Anthos Investigate Site, Passo Fundo, Rio Grande do Sul
  - Anthos Investigate Site, Porto Alegre, Rio Grande do Sul
  - Anthos Investigate Site, Marília, São Paulo
  - Anthos Investigate Site, São Paulo, São Paulo
  - Anthos Investigate Site, Votuporanga, São Paulo
- Canada (6):
  - Anthos Investigate Site, Abbotsford, British Columbia
  - Anthos Investigate Site, Newmarket, Ontario
  - Anthos Investigate Site, Oshawa, Ontario
  - Anthos Investigate Site, Toronto, Ontario
  - Anthos Investigate Site, Québec, Quebec
  - Anthos Investigate Site, Sherbrooke, Quebec
- Czechia (8):
  - Anthos Investigate Site, Jinočany, Central Bohemian
  - Anthos Investigative Site, Náchod, Hradec Králové
  - Anthos Investigative Site, Mariánské Lázně, Karlovy Vary
  - Anthos Investigative Site, Trutnov, Královéhradecký kraj
  - Anthos Investigative Site, Prague, Lekarna BENU
  - Anthos Investigative Site, Prague, Praha 5 - Hlubocepy
  - Anthos Investigate Site, Prague, Praha 5
  - Anthos Investigative Site, Ústí nad Labem, Ústí Nad Labem Region
- Germany (6):
  - Anthos Investigative Site, Obermichelbach, Bavaria
  - Anthos Investigative Site, Markkleeberg, Leipzig
  - Anthos Investigate Site, Ludwigshafen am Rhein, Ludwigshafen
  - Anthos Investigate Site, Dresden, Saxony
  - Anthos Investigative Site, Pirna, Sächsische Schweiz-Osterzgebirge
  - Anthos Investigate Site, Berlin
- Hungary (2):
  - Anthos Investigate Site, Debrecen, Hajdú-Bihar Megye
  - Anthos Investigate Site, Budapest
- Italy (8):
  - Anthos Investigate Site, Napoli, Campania
  - Anthos Investigate Site, Bergamo, Lombardy
  - Anthos Investigate Site, Milan, Lombardy
  - Anthos Investigate Site, Roma, RM
  - Anthos Investigate Site, Perugia, Umbria
  - Anthos Investigate Site, Bologna
  - Anthos Investigate Site, Sesto San Giovanni
  - Anthos Investigate Site, Varese
- Mexico (7):
  - Anthos Investigate Site, Torreón, Coahuila
  - Anthos Investigate Site, Mexico City, Cuauhtemoc
  - Anthos Investigate Site, Guadalajara, Jalisco
  - Anthos Investigate Site, San Pedro Garza García, Nuevo León
  - Anthos Investigate Site, Culiacán, Sinaloa
  - Anthos Investigate Site, Mexico City
  - Anthos Investigate Site, Querétaro
- Poland (12):
  - Anthos Investigative Site, Bochnia, Lesser Poland Voivodeship
  - Anthos Investigative Site, Lublin, Lublin Voivodeship
  - Anthos Investigate Site, Warsaw, Mazovian
  - Anthos Investigative Site, Ostrów Mazowiecka, Ostrów Mazowiecka County
  - Anthos Investigative Site, Rzeszów, Podkarpackie Voivodeship
  - Anthos Investigate Site, Bialystok, Podlaskie Voivodeship
  - Anthos Investigative Site, Bialystok, Podlaskie Voivodeship
  - Anthos Investigative Site, Czeladź, Silesian Voivodeship
  - Anthos Investigate Site, Szczecin, Zach-pomorskie
  - Anthos Investigate Site, Warsaw
  - Anthos Investigate Site, Lodz, Łódzkie Województwo
  - Anthos Investigative Site, Skierniewice, Łódź Voivodeship
- Spain (3):
  - Anthos Investigate Site, Sabadell, Barcelona
  - Anthos Investigative Site, Córdoba, Cabra
  - Anthos Investigate Site, Madrid
- United Kingdom (7):
  - Anthos Investigate Site, Peterborough, Cambridgeshite
  - Anthos Investigate Site, Hayle, Cornwall
  - Anthos Investigate Site, Norwich, Norfolk
  - Anthos Investigate Site, Ashington, Northumberland
  - Anthos Investigate Site, Newcastle, Tyne & Wear
  - Anthos Investigative Site, Barry, Vale Of Glamorgan
  - Anthos Investigate Site, Middlesex

IPD SHARING:
Plan to Share IPD: No